CLINICAL TRIAL: NCT02556931
Title: Phase II Study of Shortened-duration Tacrolimus Following Nonmyeloablative Peripheral Blood Stem Cell Transplant With High-dose Posttransplantation Cyclophosphamide in Malignancies That Are Challenging to Engraft
Brief Title: Shorter Course Tacro After NMA, Related Donor PBSCT With High-dose Posttransplant Cy for Hard-to-Engraft Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J15165; IRB00080399 (Other: JHMIRB); P01CA015396 (NIH)
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Chronic Myeloid Leukemia; Chronic Myeloproliferative Disorders; Multiple Myeloma; Plasma Cell Neoplasm; Plasma Cell Dyscrasia; Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia; Plasma Cell Leukemia
Keywords: immunosuppression; nonmyeloablative; non-myeloablative; allogeneic; tacrolimus; peripheral blood; cyclophosphamide; mycophenolate mofetil
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Paraproteinemias; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Leukemia, Plasma Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBSCT D90 (Experimental): Non-myeloablative peripheral blood stem cell transplant (PBSCT) with a fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis. Tacrolimus will be stopped at either Day 90 or Day 180 depending on GVHD status.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Drug: Tacrolimus; Drug: Mycophenolate mofetil
- PBSCT D60 (Experimental): Non-myeloablative peripheral blood stem cell transplant (PBSCT) with a fludarabine (Flu), cyclophosphamide (Cy), total body irradiation (TBI) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis. Tacrolimus will be stopped at either Day 60 or Day 180 depending on GVHD status.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Fludarabine — Days -6 through -2: 30 mg/m^2 IV daily
  Other Names: Fludara
Drug: Cyclophosphamide — Days -6 and -5: 14.5 mg/kg IV daily Days 3 and 4: 50 mg/kg IV daily
  Other Names: Cytoxan; Cy; CTX
Radiation: Total body irradiation — Day -1: 200 cGy in a single fraction
  Other Names: TBI
Drug: Tacrolimus — Start on Day 5 through either Day 60 or Day 90 depending on cohort assignment. May be continued through Day 180 depending on GVHD status.
  Other Names: Prograf; FK506; FK-506
Drug: Mycophenolate mofetil — Days 5 through 35: 15 mg/kg PO three times daily (max 3 g/day)
  Other Names: MMF; CellCept

SUMMARY:
To see if it is possible to use short-duration tacrolimus after a peripheral blood stem cell transplant in certain malignancies that are considered difficult to engraft.

DETAILED DESCRIPTION:
The main goal is to learn whether a drug called tacrolimus, which is an immune-lowering drug (an immunosuppressant) given after transplant to help prevent certain complications, can be given safely for a shorter period of time than it has been in the past. The experiences with immunosuppression duration with other allogeneic HSCT platforms cannot be directly extrapolated to the high-dose posttransplantation cyclophosphamide platform (another type of immunosuppressant given after transplant to help prevent GVHD). There are presently no published data on the minimum required duration of tacrolimus after nonmyeloablative HSCT that includes high-dose Cy as part of postgrafting immunosuppression. The effectiveness of high-dose posttransplantation Cy in GVHD prevention, however, permits the investigation of this question. At the present time there are few or no cures for diseases studied on this trial outside of a bone marrow or peripheral blood transplant. The peripheral blood for this transplant comes from a relative who is a half-match or "haplo" match to the participant. Possible donors include parents, siblings, and children. In order to help the bone marrow grow, or "take", inside the body, participants will receive chemotherapy and radiation before the transplant. After the transplant participants will receive high doses of cyclophosphamide (Cytoxan®) along with other medications to lower the immune system, such as tacrolimus. These medications may lower the risk of graft versus host disease (GVHD) and of rejection of the peripheral blood graft.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a suitable related HLA-haploidentical or -matched stem cell donor, or a 10/10 matched unrelated donor
* Eligible diagnoses: myelodysplastic syndrome (MDS) with at least 1 poor-risk feature; small lymphocytic lymphoma (SLL) or chronic lymphocytic leukemia (CLL) with 17p deletion or with progression < 6 months after a second or greater treatment regimen; T-cell prolymphocytic leukemia (PLL) in partial response or better; interferon- or tyrosine-kinase-refractory chronic myeloid leukemia (CML), or CML in second or subsequent chronic phase; Philadelphia chromosome negative (Ph-) myeloproliferative disease, including myelofibrosis; Multiple myeloma or plasma cell leukemia in partial response or better; Hematologic malignancy in complete remission with minimal residual disease (MRD) detectable by conventional cytogenetics, FISH, flow cytometry, or molecular testing
* Any previous autologous transplant must have occurred > 3 months ago
* Left ventricular ejection fraction (LVEF) >= 35%, or shortening fraction > 25%
* Bilirubin <= 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis)
* AST and ALT <= 5 x institutional upper limit of normal
* FEV1 and FVC >= 40% of predicted; if unable to perform pulmonary function testing, oxygen saturation > 92% on room air
* ECOG performance status <= 2, or Karnofsky/Lansky status >= 60

Exclusion Criteria:

* Pregnancy or active breastfeeding
* Uncontrolled active infection
* Previous allogeneic transplant
* Active extramedullary leukemia or active central nervous system (CNS) malignant disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy E DeZern, MD, Principal Investigator — 410-502-7208
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBSCT D90 | PBSCT D60
Started | 57 | 60
Completed | 57 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBSCT D90 | PBSCT D60 | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 36 | 70
  >=65 years | 23 | 24 | 47
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 78] | 63 [22 to 75] | 62.5 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 40 | 41 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 60 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Able to Stop Prophylactic Tacrolimus (D90 Cohort)
Description: This outcome measures the feasibility of stopping prophylactic tacrolimus at Day 90.
Time Frame: Day 90
Population: Safety stopping criteria were not met after discontinuation of tacrolimus at day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 57
Participants | 33

2. Primary Outcome: Percentage of Participants Who Are Able to Stop Prophylactic Tacrolimus (D60 Cohort)
Description: This outcome measures the feasibility of stopping prophylactic tacrolimus at Day 60.
Time Frame: Day 60
Population: Of the 42 patients in the D60 cohort who stopped IS early as prespecified, 10 subsequently relapsed.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 60
Participants | 42

3. Secondary Outcome: Number of Participants With Grades III-IV Acute GVHD, Days 90-180 (D90)
Description: Number of participants who experience grade III or IV acute GVHD between Day 90 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 90 are evaluable.
Time Frame: Between Day 90 and Day 180
Population: Of the 57 patients in the D90 cohort, 33 stopped tactolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 1

4. Secondary Outcome: Number of Participants With Grades III-IV Acute GVHD, Days 60-180 (D60)
Description: Number of participants who experience grade III or IV acute GVHD between Day 60 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 60 are evaluable.
Time Frame: Between Day 60 and Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 3

5. Secondary Outcome: Number of Participants With Chronic GVHD, Days 90-180 (D90)
Description: Number of participants who experience chronic GVHD requiring additional immunosuppressive therapy between Day 90 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 90 are evaluable.
Time Frame: Between Day 90 and Day 180
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 2

6. Secondary Outcome: Number of Participants With Chronic GVHD, Days 60-180 (D60)
Description: Number of participants who experience chronic GVHD requiring additional immunosuppressive therapy between Day 60 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 60 are evaluable.
Time Frame: Between Day 60 and Day 180
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 1

7. Secondary Outcome: Number of Participants Who Experience Graft Failure, Days 90-180 (D90)
Description: Number of participants who experience graft failure between Day 90 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 90 are evaluable.
Time Frame: Between Day 90 and Day 180
Population: Of the 57 patients in the D90 cohort, 33 stopped IS early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 0

8. Secondary Outcome: Number of Participants Who Experience Graft Failure, Days 60-180 (D60)
Description: Number of participants who experience graft failure between Day 60 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 60 are evaluable.
Time Frame: Between Day 60 and Day 180
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 1

9. Secondary Outcome: Number of Participants Who Experience Disease Relapse, Days 90-180 (D90)
Description: Number of participants who experience disease relapse between Day 90 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 90 are evaluable.
Time Frame: Between Day 90 and Day 180
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 14

10. Secondary Outcome: Number of Participants Who Experience Disease Relapse, Days 60-180 (D60)
Description: Number of participants who experience disease relapse between Day 60 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 60 are evaluable.
Time Frame: Between Day 60 and Day 180
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 10

11. Secondary Outcome: Number of Participants Who Experience Non-relapse Mortality, Days 90-180 (D90)
Description: Number of participants who die for any reason other than disease relapse between Day 90 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 90 are evaluable.
Time Frame: Between Day 90 and Day 180
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 1

12. Secondary Outcome: Number of Participants Who Experience Non-relapse Mortality, Days 60-180 (D60)
Description: Number of participants who die for any reason other than disease relapse between Day 60 and Day 180. Only participants who are able to stop prophylactic tacrolimus at Day 60 are evaluable.
Time Frame: Between Day 60 and Day 180
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 2

13. Secondary Outcome: Number of Participants Who Experience Grades III-IV GVHD, Day 360 (D90)
Description: Number of participants who experience grade III or IV GVHD by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 16

14. Secondary Outcome: Number of Number of Participants Who Experience Grades III-IV GVHD, Day 360 (D60)
Description: Number of participants who experience grade III or IV GVHD by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 18

15. Secondary Outcome: Number of Number of Participants With Severe Chronic GVHD, Day 360 (D90)
Description: Number of participants who experience severe chronic GVHD requiring additional immunosuppressive therapy by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 7

16. Secondary Outcome: Number of Number of Participants With Severe Chronic GVHD, Day 360 (D60)
Description: as for outcome 15
Time Frame: Day 360
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 5

17. Secondary Outcome: Number of Number of Participants Who Experience Graft Failure, Day 360 (D90)
Description: Number of participants who experience graft failure by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 0

18. Secondary Outcome: Number of Number of Participants Who Experience Graft Failure, Day 360 (D60)
Description: Number of participants who experience graft failure by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 2

19. Secondary Outcome: Number of Participants Who Experience Relapse, Day 360 (D90)
Description: Number of participants who experience disease relapse by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 14

20. Secondary Outcome: Number of Participants Who Experience Relapse, Day 360 (D60)
Description: Number of participants who experience disease relapse by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 10

21. Secondary Outcome: Number of Participants Who Experience Non-relapse Mortality, Day 360 (D90)
Description: Number of participants who die for any reason other than disease relapse by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 57 patients in the D90 cohort, 33 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D90
Number analyzed (Participants) | 33
Participants | 4

22. Secondary Outcome: Number of Participants Who Experience Non-relapse Mortality, Day 360 (D60)
Description: Number of participants who die for any reason other than disease relapse by Day 360. All participants are evaluable.
Time Frame: Day 360
Population: Of the 60 patients in the D60 cohort, 42 stopped tacrolimus early as planned.
Measure: Count of Participants; unit: Participants
Arm/Group | PBSCT D60
Number analyzed (Participants) | 42
Participants | 4

ADVERSE EVENTS:
Time Frame: adverse event data were collected for each particpant for at minimum 1 year. Median follow-up of 41 months in the D90 cohort and 27 months in the D60 cohort.
Arm/Group | PBSCT D90 | PBSCT D60
All-Cause Mortality (participants affected / at risk) | 12/57 | 10/60
Serious Adverse Events (participants affected / at risk) | 9/57 | 5/60
Other Adverse Events (participants affected / at risk) | 35/57 | 16/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBSCT D90 (N=57) | PBSCT D60 (N=60)
Severe cGVHD (Skin and subcutaneous tissue disorders) | 9 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBSCT D90 (N=57) | PBSCT D60 (N=60)
neutropenic fever (Infections and infestations) | 35 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02556931/Prot_SAP_000.pdf